CLINICAL TRIAL: NCT02489370
Title: CHF Home Telemonitoring: A Home Telemonitoring Service for Chronic Heart Failure Patients on Trial
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital of North Norway (Other)
Responsible Party: Principal Investigator, Artur Serrano, Senior Research Scientist, University Hospital of North Norway
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2013/356/REK nord
Record Dates: First submitted 2015-06-25; First posted 2015-07-03 (Estimated); Last update posted 2015-07-03 (Estimated); Status verified 2015-07

CONDITIONS: Congestive Heart Failure
Keywords: home care; telecare; telehealth; telemonitoring; chronic heart failure; randomized controlled trial; Congestive Heart Failure; telemedicine
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Telemonitoring (intervention) (Experimental): an intervention arm testing the proposed telemonitoring service and a control arm with the current treatment.
  Patients assigned to the intervention arm receive a home telemonitoring kit consisting of a tablet, a wireless weight scale and a portable blood pressure meter. The patient is asked to weigh him- or herself every day and the monitoring procedure happens as previously described. In addition a measurement of the blood pressure is also made.
  Interventions: Device: Home telemonitoring
- Usual care (control) (No Intervention): Patients assigned to the control arm receive treatment as usual, consisting of a recommendation to weigh themselves at home, using their own weight scale, and to report by phone to the polyclinic if there is a significant change in weight.

INTERVENTIONS:
Device: Home telemonitoring — The intervention consists of daily monitoring the patients' weight and blood pressure directly from their home; automatically and securely transmit the values to a server at the hospital; and monitor the values by a trained nurse at the Heart polyclinic.
  Other Names: Telecare; Telehealth
  Arms: Telemonitoring (intervention)

SUMMARY:
Providing patients with chronic heart failure (CHF) access to remote monitoring, for example by telephone or telemonitoring using wireless technology, reduces deaths and hospitalisations and may provide benefits on health care costs and quality of life. Remote monitoring of patients with chronic heart failure can reduce pressure on resources, particularly for conditions like chronic heart failure, which exert a large burden on health services. These are conclusions of the Cochrane Systematic Review from 2010.

In Norway the costs for treatment of chronic heart failure are vast, both concerning hospital treatment, daily use of medication over years, and loss of quality of life for patients and their family caregivers. Generally there is little knowledge about what is gained for the billions used. In Norway no telemonitoring services are established and hence no investigations have yet been published. Thus it seems that current evidence of effectiveness and quality is insufficient to recommend usage. The structure and funding streams in Norwegian health services are different from other countries and the conventional services that the intervention has been compared to in previous studies, are most likely heterogeneous. It is thus important to investigate Norwegian conditions.

Advanced telemonitoring technology with electronic transfer of physiological data such as blood pressure and weight is currently being used in research and established routine services in several countries in Europe, amongst them the Netherlands, Germany and the United Kingdom.

The proposed project intends to introduce such a strategy as an avenue for exploring promising new services that would not otherwise be available in Norway. The service consists of daily monitoring the patients' weight and blood pressure directly from their home; automatically and securely transmit the values to a server at the University Hospital of North Norway (UNN); and monitor the values by a trained nurse at the Heart polyclinic.

The primary objective of this study is thus to explore whether, as compared to current care from the Heart Polyclinic, the introduction of home telemonitoring will reduce hospital readmissions and will, in addition, be cost-effective. This is in line with current directions of European telemonitoring programmes for patients with chronic heart failure. This result may define if the telemonitoring of heart failure patients is feasible for Norway or not at all.

DETAILED DESCRIPTION:
All data collected by the equipment placed at the patient's home will be directly and securely transferred to the Heart polyclinic of the University Hospital of North Norway (UNN). All data is anonymous as explained below, only the weight and the codes with the answers to the questionnaire are send.

Each day a nurse is assigned as responsible for the heart remote monitoring system. The nurse in charge must read the heart remote monitoring email in the morning every day, seven days a week. If an alert email has been received, then the nurse logs into the system's dashboard and reads the data displayed there for that patient. Then the nurse will try to phone the patient to clarify the situation. Until this moment the procedure protocol differs from the ordinary routines as the notification of a case is usually raised by a phone call from the patient or a hospitalisation. But from this moment on, the procedure protocol is the same as for all patients treated by the Heart polyclinic, i.e. if the nurse evaluates the situation to need a further follow-up, then the nurse contacts the patient's general practitioner (GP) by phone (as said this is procedure as usual). The hospital's Heart polyclinic has the same responsibility for the treatment of the patients, both in the intervention arm and the control arm.

Each one of the patients assigned to the intervention arm will be following this procedure during 6 months. For the patients assigned to the control arm they will receive treatment as usual also during a period of 6 months. Data stored in the system is anonymised. All patients are uniquely identified by a number, the Unique Identifier (UID), in the system, the connection between the UID and the real identity being only stored in a file in a secured personal computer unconnected from any network, staying in an office at the heart polyclinic. Once a week, the UIDs' file stored in the study personal computer at the Heart polyclinic is transferred to a hardware protected pen drive. The pen drive in then placed in another building at the UNN. This procedure is of the responsibility of the UNN's department for "E-health and information and communications technology (ICT)". In this way only two copies of the file are stored in separate buildings. No reference to the study name is mentioned in this file.

As a pilot study, a prototype of the platform was built. It consisted of a wireless weight scale and also a blood pressure meter prepared to send the values through the home Wi-Fi network to a connected portable computer. The portable computer could then send the encrypted measurements to a server at UNN.

After the first two months of pilot testing, the patient was satisfied with the usability of the solution and the reliability of the service was proven.

The platform deployed and tested in the pilot study has been extended to include functionalities for multiple patients. A dashboard showing all the measurements received (unidentified) has been developed for the polyclinic and used by the responsible clinician (the nurse on daily duty). This data is unidentified and consists of a registration of blood pressure and weight, the encoded answers to the questionnaire attached (example: Q3A2 means that question 3 got the answer 2 in the questionnaire). The responsible nurse at the Heart Polyclinic has access to the dashboard. When a situation requiring the nurse intervention arises, the system sends an alerting email to a pre-defined address (usually the nurse's email account as it will be done in this study).

The design of the randomized controlled trial (RCT) Power analysis The inclusion of 40 patients is based upon the total number of new patients served by the polyclinic per year during the 2 last years. For this study a sample size was calculated based on a readmission rate of 70% of the patients per year on average with a standard deviation of 20pp (percentage points). The values are adequate, based on patients who have received treatment within the Heart Polyclinic and also replicating the study by Antonicelli, published in the Journal of telemedicine and Telecare "Impact of telemonitoring at home on the management of elderly patients with congestive heart failure" in 2008.

It was assumed by the clinical team that a 1/3 reduction on the rate of readmissions (down to 47%) would be clinically relevant as the margin of superiority for the intervention. To have 95% certainty (power) that a test at 0.05 level of significance would find a statistically significant difference between the means, the study would include a minimum of 20 patients in each group.

The planned RCT The telemonitoring service will be offered to all patients admitted at UNN's Heart Polyclinic, satisfying the inclusion criteria. The study comprises an intervention arm testing the proposed telemonitoring service and a control arm with the current treatment.

Patients assigned to the intervention arm receive a home telemonitoring kit consisting of a tablet, a wireless weight scale and a portable blood pressure meter. The patient is asked to weigh him- or herself every day and the monitoring procedure happens as previously described. In addition a measurement of the blood pressure is also made.

Patients assigned to the control arm receive treatment as usual, consisting of a recommendation to weigh themselves at home, using their own weight scale, and to report by phone to the polyclinic if there is a significant change in weight.

The study calendar is shown below. Recruiting period: 14 months Follow-up period: 6 months Number of patients: 40

Randomization: will be performed using sequentially numbered sealed opaque envelopes

Blinding: independent outcome assessors and data analysts are blinded to which group the patient has been assigned to (patients are not blinded due to the nature of the intervention).

Challenges and opportunities Qualitative research with semi structured interviews. Patients in the intervention group and health care professionals will be asked to state their opinion of the service. The research team will also observe patients' interactions with the system after the 6 months of the study. A qualitative summary and thematic analysis of significant features of opinions and actions will be connected to best practices. The purpose is to be able to understand how best practices can be developed in the Northern Norwegian context, and describe their mechanisms. The innovation intention is to adjust the services as they develop, by considering the identified additional conditions for future development.

Ethics and privacy With recent events and advances in information technology and the Internet, confidentiality regarding handling of patient private data has become a critical aspect of a study design as privacy is a fundamental right in the public healthcare domain. In this project confidentiality of private health information will be ensured according to the Health Personnel Act § 21, helsepersonelloven § 21, and described in LOV2001-05-18 nr.24 (Helse- og omsorgsdepartementet, 2001). All private personal data will be de-identified: every unique identifying number, characteristic, or code identifiers of the individual or of relatives, employers, or household members of the individual will be removed so that the information can be used alone or in combination with other information. The resulting data will be analysed by a statistician to ensure that no individually identifiable health information remains. The consent of participants will be required by means of providing a letter of informed consent to be signed.

ELIGIBILITY:
Inclusion Criteria:

Presence of CHF signs and symptoms such as dyspnoea and peripheral or pulmonary oedema requiring diuretic administration (New York Heart Association [NYHA] functional class II-IV); and ejection fraction (EF) under 40% combined or not with a left ventricular filling pattern supporting the presence of diastolic dysfunction, according to the American College of Cardiology/American Heart Association Guidelines for chronic heart failure.

Exclusion Criteria:

Severe psychiatric disturbance diagnosed by DSM-IV-TR criteria. Any disability that may prevent the subject from completing the informed consent form or other study requirements.

Medication or drug dependency or abuse (except for nicotine). Inability to handle the technological devices included in the study, for some other reason.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2014-10; Primary Completion 2016-06 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Heart failure related hospital readmissions | Intervention period (6 months)
  Calculated as the proportion of patients readmitted to hospital at least once during the period of follow-up
Additional costs/savings resulting from the service | 6 months
  Defined as the difference in the costs of medical care during the study, identified through a cost analysis, between the intervention and control arms

SECONDARY OUTCOMES:
Length of stay | 6 months
  Defined as the length of stay per hospitalization
Assessment of Quality of Life | At baseline and end of study (6 months)
  Based on the Minnesota Living with Heart Failure questionnaire (MLWHF)

CONTACTS AND LOCATIONS:
Overall Officials: J. Artur Serrano, PhD, Principal Investigator — Senior Research Scientist, Norwegian Centre for Telemedicine, University Hospital of North Norway; Paal Tande, MD, Study Director — Leader Cardiology Department, University Hospital of North Norway; Marina Nilsen, Nurse, Study Chair — Leader Heart Polyclinic, University Hospital of North Norway
Locations (1):
- University Hospital of North Norway, Tromsø, Troms, Norway